CLINICAL TRIAL: NCT01472757
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Study to Evaluate the Efficacy and Safety of VR506 Inhaled From a New Inhaler in Adolescent and Adult Subjects With Asthma
Brief Title: Clinical Study to Evaluate the Efficacy of VR506 Using a New Inhaler for the Treatment of Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VR506/2/002
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 1 (Active Comparator)
  Interventions: Drug: VR506
- Dose 2 (Active Comparator)
  Interventions: Drug: VR506
- Dose 3 (Active Comparator)
  Interventions: Drug: VR506

INTERVENTIONS:
Drug: VR506 — VR506 inhalation powder delivered via a new dry powder inhaler
  Arms: Dose 1; Dose 2; Dose 3
Drug: Placebo — Placebo delivered via a new dry powder inhaler
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the clinical efficacy of three doses of VR506 delivered via a new dry powder inhaler for the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adolescents aged 12 to 17 years (inclusive) and adults aged 18 to 65 years (inclusive)
* Documented clinical history of asthma (i.e. made by a physician) for at least 6 months before the Screening Visit
* Documented asthma reversibility in the 5 years prior to or during Screening, or if the asthma reversibility criterion is not met at Screening, then a repeat test may be carried out at the end of the Run-In Period
* Subjects with asthma who, in the opinion of the investigator, require maintenance therapy with inhaled corticosteroids (ICS), are believed to have been regularly compliant with this therapy, and are therefore likely to deteriorate within 6 weeks following withdrawal of their usual ICS treatment
* Mild or moderate asthma, defined as:

  * Mild - good asthma control achieved by low-dose inhaled corticosteroid (daily dose 200-500 μg beclomethasone dipropionate or equivalent) with or without other low-intensity treatment (e.g. leukotriene modifiers or cromones) for at least 28 days before the Screening Visit
  * Moderate - good asthma control achieved by low- to moderate-dose ICS (daily dose 200-1000 μg beclomethasone dipropionate or equivalent), and long acting β2-agonist (LABA) or other extra treatment, for at least 28 days before the Screening Visit
* Ability to use the new inhaler correctly, based on investigator's review of the completed inhaler operation checklist
* Ability to use the eDiary correctly, assessed by the investigator during the Screening Period
* Ability to perform technically satisfactory pulmonary function tests
* Ability to comply with study procedures, including blood sampling
* Body mass index (BMI) of 16.0 to 26.0 kg/m2 in adolescents, and in adult subjects recruited in the Philippines, and 18.0 to 32.0 kg/m2 in adults recruited in other countries
* Available to complete all study visits
* Oral peak inspiratory flow (PIF) of at least 60 L/min; using an appropriate device set to match the resistance of the new dry powder inhaler (nDPI)
* Good health, except for the presence of asthma, according to medical history and physical examination
* Normal (i.e. non-clinically significant abnormality) 12-lead electrocardiogram (ECG)
* Negative drug, alcohol, and urine cotinine screen; subjects must test negative for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, cotinine (unless related to nicotine-containing therapies), ethanol, and opiates (unless given as a prescription medicine)
* Non-smokers or ex-smokers with a smoking history of less than 10 pack-years (e.g. <20 cigarettes per day for 10 years or 40 cigarettes per day for 5 years) and stopped smoking for at least one year prior to the Screening Visit. Smoking will not be permitted throughout the study
* Female subjects of child-bearing potential must be using medically acceptable forms of contraception; approved forms of contraception are abstinence, hormonal (oral, implant, transdermal, or injection, in use for ≥3 consecutive months before the start of the Run-In Period), double barrier (condom with spermicide, diaphragm with spermicide), intrauterine device, or vasectomised partner (≥6 months since vasectomy)

Exclusion Criteria:

* Regular use (≥3 times per week) of topical steroids taken to treat dermatitis, rhinitis or allergic conjunctivitis, within 28 days of the Screening Visit
* Subjects who have or who have had an upper or lower respiratory tract infection within 28 days of the Screening Visit
* Subjects with asthma that required admission to an intensive care unit and/or ventilation within the previous 12 months
* History of lung cancer
* Subjects with "brittle asthma", defined as patients with asthma who either maintain over many months a wide variation (>40%) in peak expiratory flow (PEF) between morning and evening measurements despite moderate to high doses of ICS, or are prone to acute, severe and often unpredictable attacks of asthma that may be fatal, on a background of apparently good asthma control
* History or current diagnosis of human immunodeficiency virus (HIV) infection
* Active chronic hepatitis B or C infection. If the patient's screening test is positive for hepatitis B surface antigen, the patient should be excluded unless the investigator, after a careful review of the patient's medical history and current laboratory tests of liver function, can exclude the possibility of recent or current infection
* Persistent arterial hypotension, with average systolic blood pressure (SBP) readings of ≤95 mmHg
* Subjects who have any clinically significant abnormality or finding from examination, tests, or history that may compromise subject safety, specifically any history of cardiac, renal or hepatic impairment
* Subjects with an abnormal ECG
* Persistent elevation of blood pressure, with average SBP readings of ≥160 mmHg or average diastolic blood pressure (DBP) readings of ≥100 mmHg
* Pregnant or lactating females
* Participation in another clinical study in the 28 days prior to the Screening Visit
* Current or a history of drug or alcohol abuse or dependence according to World Health Organization criteria in the 12 months prior to the Screening Visit or evidence of such abuse as indicated by laboratory assays conducted during the screening evaluation
* Evidence of clinically significant renal, hepatic, cardiac, pulmonary (apart from asthma) or metabolic dysfunction, e.g. diabetes mellitus, thyrotoxicosis, uncorrected hypokalaemia, or predisposition to low levels of serum potassium
* Inability to communicate well with the investigator
* Evidence of clinically significant renal, hepatic, cardiac, pulmonary (apart from asthma) or metabolic dysfunction, e.g. diabetes mellitus, thyrotoxicosis, uncorrected hypokalaemia, or predisposition to low levels of serum potassium
* Donation of ≥450 mL of blood or blood products within the previous 12 weeks prior to the Screening Visit
* History of allergy, intolerance or contraindications to corticosteroids, lactose, or severe allergy to milk proteins
* Consumption of alcohol- or caffeine-containing foods or beverages from midnight before or during the Screening Visit. The visit can be rescheduled once before the subject is excluded
* History of medically diagnosed chronic respiratory diseases (other than asthma) e.g. chronic obstructive pulmonary disease
* Subjects with previously clinically or radiologically diagnosed osteoporosis and/or those receiving regular treatment (more than 1 month duration) with oral or parenteral corticosteroids in the last year prior to the Screening Visit

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Dr., Principal Investigator — Aarhus University Hospital
Locations (82):
- United States (32):
  - Vectura Clinical Trial Site 10038, Fountain Valley, California
  - Vectura Clinical Trial Site 10031, Los Angeles, California
  - Vectura Clinical Trial Site 10044, Mission Viejo, California
  - Vectura Clinical Trial Site 10022, Orange, California
  - Vectura Clinical Trial Site 10014, Rancho Mirage, California
  - Vectura Clinical Trial Site 10027, Rolling Hills Estates, California
  - Vectura Clinical Trial Site 10033, San Jose, California
  - Vectura Clinical Trial Site 10016, Vista, California
  - Vectura Clinical Trial Site 10023, Centennial, Colorado
  - Vectura Clinical Trial Site 10001, Colorado Springs, Colorado
  - Vectura Clinical Trial Site 10025, Denver, Colorado
  - Vectura Clinical Trial Site 10041, Sarasota, Florida
  - Vectura Clinical Trial Site 10011, Albany, Georgia
  - Vectura Clinical Trial Site 10002, Metairie, Louisiana
  - Vectura Clinical Trial Site 10042, Baltimore, Maryland
  - Vectura Clinical Trial Site 10029, North Dartmouth, Massachusetts
  - Vectura Clinical Trial Site 10008, Plymouth, Minnesota
  - Vectura Clinical Trial Site 10020, Warrensburg, Missouri
  - Vectura Clinical Trial Site 10009, Missoula, Montana
  - Vectura Clinical Trial Site 10034, Bellevue, Nebraska
  - Vectura Clinical Trial Site 10035, Omaha, Nebraska
  - Vectura Clinical Trial Site 10015, Omaha, Nebraska
  - Vectura Clinical Trial Site 10040, Rochester, New York
  - Vectura Clinical Trial Site 10010, Sylvania, Ohio
  - Vectura Clinical Trial Site 10017, Oklahoma City, Oklahoma
  - Vectura Clinical Trial Site 10028, Medford, Oregon
  - Vectura Clinical Trial Site 10024, Portland, Oregon
  - Vectura Clinical Trial Site 10021, Upland, Pennsylvania
  - Vectura Clinical Trial Site 10003, Charleston, South Carolina
  - Vectura Clinical Trial Site 10019, Boerne, Texas
  - Vectura Clinical Trial Site 10039, Waco, Texas
  - Vectura Clinical Trial Site 10004, Draper, Utah
- Philippines (6):
  - Vectura Clinical Trial Site 31001, Lipa City, Batangas
  - Vectura Clinical Trial Site 31002, Davao City
  - Vectura Clinical Trial Site 31003, Iloilo City
  - Vectura Clinical Trial Site 31004, Pasig
  - Vectura Clinical Trial Site 31005, Quezon City
  - Vectura Clinical Trial Site 31007, Quezon City
- Poland (16):
  - Vectura Clinical Trial Site 20018, Bialystok
  - Vectura Clinical Trial Site 20013, Biołystok
  - Vectura Clinical Trial Site 20015, Krakow
  - Vectura Clinical Trial Site 20019, Krakow
  - Vectura Clinical Trial Site 20009, Lodz
  - Vectura Clinical Trial Site 20012, Lublin
  - Vectura Clinical Trial Site 20008, Ostrów Wielkopolski
  - Vectura Clinical Trial Site 20003, Poznan
  - Vectura Clinical Trial Site 20005, Poznan
  - Vectura Clinical Trial Site 20016, Skiemiewice
  - Vectura Clinical Trial Site 20021, Tarnów
  - Vectura Clinical Trial Site 20010, Warsaw
  - Vectura Clinical Trial Site 20001, Wroclaw
  - Vectura Clinical Trial Site 20006, Wroclaw
  - Vectura Clinical Trial Site 20014, Zawadzkie
  - Vectura Clinical Trial Site 20007, Łodź
- Romania (11):
  - Vectura Clinical Trial Site 21002, Brasov
  - Vectura Clinical Trial Site 21011, Bucharest
  - Vectura Clinical Trial Site 21004, Cluj-Napoca
  - Vectura Clinical Trial Site 21009, Cluj-Napoca
  - Vectura Clinical Trial Site 21010, Cluj-Napoca
  - Vectura Clinical Trial Site 21007, Iași
  - Vectura Clinical Trial Site 21008, Iași
  - Vectura Clinical Trial Site 21013, Judetul Cluj
  - Vectura Clinical Trial Site 21012, Judetul Iasi
  - Vectura Clinical Trial Site 21001, Târgu Mureş
  - Vectura Clinical Trial Site 21005, Timișoara
- Ukraine (17):
  - Vectura Clinical Trial Site 23013, Donetsk
  - Vectura Clinical Trial Site 23005, Kharkiv
  - Vectura Clinical Trial Site 23004, Kharkiv
  - Vectura Clinical Trial Site 23010, Kharkiv
  - Vectura Clinical Trial Site 23012, Kiev
  - Vectura Clinical Trial Site 23002, Kiev
  - Vectura Clinical Trial Site 23009, Kiev
  - Vectura Clinical Trial Site 23011, Kiev
  - Vectura Clinical Trial Site 23017, Kiev
  - Vectura Clinical Trial Site 23001, Kyiv
  - Vectura Clinical Trial Site 23003, Kyiv
  - Vectura Clinical Trial Site 23018, Kyiv
  - Vectura Clinical Trial Site 23007, Odesa
  - Vectura Clinical Trial Site 23015, Simferopol
  - Vectura Clinical Trial Site 23014, Vinnytsia
  - Vectura Clinical Trial Site 23008, Zaporizhzhya
  - Vectura Clinical Trial Site 23016, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 374 subjects were randomised, and 373 received at least one dose of study drug; 1 subject was randomised but not treated.
Groups:
- VR506 50 mcg: VR506 50 mcg inhalation powder delivered via a new dry powder inhaler
- VR506 100 mcg: VR506 100 mcg inhalation powder delivered via a new dry powder inhaler
- VR506 250 mcg: VR506 250 mcg inhalation powder delivered via a new dry powder inhaler
Period: Overall Study
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
Started | 91 | 93 | 95 | 94
Full Analysis Set (Five subjects had no post-dose efficacy assessments and were excluded from the Full Analysis Set.) | 91 | 93 | 92 | 92
Completed | 61 | 80 | 76 | 75
Not Completed | 30 | 13 | 19 | 19
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 0
Not completed — Asthma exacerbation | 4 | 1 | 2 | 1
Not completed — Treatment period withdrawal criteria met | 21 | 8 | 9 | 12
Not completed — Protocol Violation | 3 | 2 | 4 | 4
Not completed — Other reasons | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg | Total
Number analyzed (Participants) | 91 | 93 | 95 | 94 | 373
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 12 | 14 | 54
  Between 18 and 65 years | 77 | 79 | 83 | 80 | 319
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (16.2) | 38.8 (16.1) | 39.8 (15.6) | 39.3 (15.3) | 39.5 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 50 | 61 | 58 | 226
  Male | 34 | 43 | 34 | 36 | 147
Region of Enrollment [Number; unit: participants]
  Romania | 4 | 5 | 6 | 4 | 19
  United States | 18 | 19 | 19 | 19 | 75
  Philippines | 24 | 22 | 24 | 21 | 91
  Ukraine | 22 | 22 | 22 | 24 | 90
  Poland | 23 | 25 | 24 | 26 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 12) for In-clinic Morning Pre-Dose Forced Expiratory Volume In 1 Second (FEV1)
Time Frame: Baseline and 12 weeks
Population: Full analysis set analyzed, but number of patients represents subjects with both start of treatment baseline value and end of treatment value where a Last Observation Carried Forward (LOCF) approach was used to impute values of missing post-baseline visits; 2 subjects had no post-dose FEV1 assessments, baseline values were not carried forward
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
Number analyzed (Participants) | 90 | 93 | 92 | 91
Liters | 0.19 (0.36) | 0.32 (0.46) | 0.38 (0.30) | 0.38 (0.33)
Statistical Analysis 1: Comparison: Placebo vs VR506 50 mcg; Test type: Superiority; p = 0.013, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VR506 100 mcg; Test type: Superiority; p < 0.001, ANCOVA — Calculated p-value was less than 0.001
Statistical Analysis 3: Comparison: Placebo vs VR506 250 mcg; Test type: Superiority; p < 0.001, ANCOVA — Calculated p-value was less than 0.001

2. Secondary Outcome: Number of Participants With Withdrawals Due to Worsening of Asthma
Time Frame: 12 weeks
Population: Number of participants analyzed aligns with Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
Number analyzed (Participants) | 91 | 93 | 92 | 92
Participants | 26 | 9 | 11 | 12
Statistical Analysis 1: Comparison: Placebo vs VR506 50 mcg; Test type: Superiority; p = 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs VR506 100 mcg; Test type: Superiority; p = 0.006, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs VR506 250 mcg; Test type: Superiority; p = 0.011, Fisher Exact

3. Secondary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 12) for In-clinic Weekly Morning Pre-dose Peak Expiratory Flow (PEF)
Time Frame: Baseline and 12 weeks
Population: Full Analysis Set analyzed, but number of patients analyzed represents subjects with both start of treatment baseline value and end of treatment value where a Last Observation Carried Forward (LOCF) approach was used to impute values of missing post-baseline visits; 1 subject had no post-dose PEF assessment, baseline values were not carried forward
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
Number analyzed (Participants) | 90 | 93 | 92 | 92
L/min | 1.18 (47.54) | 25.00 (58.33) | 27.11 (56.67) | 21.99 (45.03)
Statistical Analysis 1: Comparison: Placebo vs VR506 50 mcg; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs VR506 100 mcg; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs VR506 250 mcg; Test type: Superiority; p = 0.008, ANCOVA

4. Secondary Outcome: Assessment of Acceptability of the Device
Description: Percentage of subjects that overall found it very easy, fairly easy or fairy difficult to use the inhaler, based on inhaler acceptability questionnaire.
Time Frame: 12 weeks
Population: Number of participants analyzed aligns with Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
Number analyzed (Participants) | 91 | 93 | 92 | 92
Participants
  Very Easy | 57 | 66 | 58 | 59
  Fairly Easy | 20 | 25 | 26 | 22
  Fairly Difficult | 2 | 0 | 0 | 2
  Missing | 12 | 2 | 8 | 9

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | VR506 50 mcg | VR506 100 mcg | VR506 250 mcg
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/93 | 0/95 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/93 | 1/95 | 0/94
Other Adverse Events (participants affected / at risk) | 47/91 | 42/93 | 40/95 | 33/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | VR506 50 mcg (N=93) | VR506 100 mcg (N=95) | VR506 250 mcg (N=94)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | VR506 50 mcg (N=93) | VR506 100 mcg (N=95) | VR506 250 mcg (N=94)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 16 (18) | 16 (17) | 12 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALLERGIC COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SPUTUM RETENTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 8 (8) | 2 (2) | 3 (4) | 2 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 5 (6) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
PHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ACUTE TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DENGUE FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRACHEITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 4 (5) | 3 (3) | 4 (4)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GASTRODUODENITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GINGIVITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GALLBLADDER PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication can be delayed for 60 days for Sponsor review and revisions/deletions can be required. Furthermore, a 6-month delay to publication can be required by the Sponsor in order to take steps to protect its proprietary information and/or intellectual property rights.